CLINICAL TRIAL: NCT02269592
Title: Study of Precursor Hematological Malignancies to Assess the Relationship Between Molecular Events of Progression and Clinical Outcome
Brief Title: Study of MGUS, Smoldering Myeloma, Early MDS and CLL to Assess Molecular Events of Progression and Clinical Outcome
Status: Recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 14-174
Record Dates: First submitted 2014-10-09; First posted 2014-10-21 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance (MGUS); Myelodysplastic Syndromes; Hematological Malignancies; B-cell Malignancy, Low-grade; Myelodysplastic Syndrome With Low-grade Lesions; IgG Monoclonal Gammopathy of Uncertain Significance; Smoldering Multiple Myeloma; Waldenstrom Macroglobulinemia
Keywords: MGUS; Smoldering Myeloma; Acute Myeloid Leukemia; Waldenstrom Macroglobulinemia; Monoclonal Gammopathy of Undermined Significance; Monoclonal B cell lymphocytosis; Smoldering Multiple Myeloma; Myelodysplastic syndromes
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Myelodysplastic Syndromes; Hematologic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Smoldering Multiple Myeloma; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, bone marrow, buccal swabs or mouthwashes, urine, lymph node biopsies, stool, discarded tissue or other specimens.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Specimen Collection: Patients' tumor tissue including bone marrow, blood, buccal swab or mouthwash, lymph node, urine or other specimens will be collected from patients who consent to the protocol

SUMMARY:
Blood cancers occur when the molecules that control normal cell growth are damaged. Many of these changes can be detected by directly examining parts of the cancer or cells in blood. Several alterations that occur repeatedly in certain types of blood cancers have already been identified, and these discoveries have led to the development of new drugs that target those alterations. More remain to be discovered.

Some of these abnormalities include alterations in genes. Genes are the part of cells that contain the instructions which tell the investigators bodies how to grow and work, and determine physical characteristics such as hair and eye color. Genes are composed of DNA letters that spell out these instructions. Studies of the DNA molecules that make up the genes are called "molecular" analyses. Molecular analyses are ways of reading the DNA letters to identify errors in genes that may contribute to an increased risk of cancer or to the behavior of the cancer cells. Some changes in genes occur only in cancer cells. Others occur in the genes that are passed from parent to child. This research study will examine both kinds of genes. The best way to find these genes is to study large numbers of people. The investigators expect that as many 1000 individuals will enroll in this study.

This research study is trying to help doctors and scientists understand why cancer occurs and to develop ways to better treat and prevent it. To participate in this study the participant must have cancer now, had it in the past, or are at risk of developing cancer. The participant will not undergo tests or procedures that are not required as part of their routine clinical care. The investigators will ask the participant to provide an additional sample from tissue that is obtained for their clinical care including blood, bone marrow, or tissue sample. The investigators will also ask for a gentle scrape of the inside of their cheek, mouthwash or a skin sample to obtain their germline DNA

DETAILED DESCRIPTION:
The purpose of this research study is to perform these molecular analyses on tissues (obtained from biopsies), blood, or other body fluids such as saliva. Importantly, this study will use tissue specimens that have already been collected as part of a participant's clinical care. The participant's tissue sample may be used to create a living tissue sample (called a "cell line") that can be grown in the laboratory. This allows researchers to have an unlimited supply of cells in the future without asking for more samples.

In this study, analyses will be performed on material only after all necessary clinical tests have been performed. In general, no additional procedures will be required. However, the investigators are asking the participant's permission to obtain one additional sample of blood (a few teaspoons), a gentle swab from the inside of their mouth or a sample of skin to obtain some cells. These are sources of normal, non-cancer cells which are needed for some types of analyses.

To fully understand the effects that molecular alterations have on blood cancers, they must be analyzed in the context of clinical behavior. Therefore, this study also asks the participant's permission to link the molecular alterations in their cancer or leukemia with clinical information that has been generated during the course of their clinical care. No additional clinical tests will be required. The investigator will ask to see the participant for follow up at regular interval to follow their risk of progression.

Some of participant's specimens as well as some of the material generated during the analysis of their tissues or blood may be useful for future study. The Investigator's are asking for the participant's permission to store these specimens and materials in a secure storage facility for possible later use.

Finally, rapid progress in understanding and treating cancer will occur when some of the molecular information derived from tissue and blood can be shared with other researchers. In particular, the National Institutes of Health (NIH) and other organizations have developed special data (information) repositories that analyze data and collect the results of certain types of genetic studies. These central banks will store genetic information and samples and give them to other researchers to do more studies. Therefore, the Investigators are also asking your permission to share your results with these special banks. The participant's information will be sent with only a code number attached. The participant's name or other directly identifiable information will not be given to central banks. There are many safeguards in place to protect the participant's information and samples while stored in repositories and used for research. The investigators do not think that there will be further risks to the participant's privacy and confidentiality by sharing this information with these banks. However, the investigator's cannot predict how genetic information will be used in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Known or Suspected Precursor Hematological Cancer
* Including the following subgroups of diseases:

  * Early MDS, including pathologically-confirmed MDS (IPSS Low/Int-1; IPSS-R Very Low/Low) and idiopathic cytopenias of undetermined significance (ICUS);
  * Asymptomatic Multiple Myeloma and Waldenstrom Macroglobulinemia such as monoclonal gammopathy of undermined significance (MGUS) or Smoldering Multiple Myeloma (SMM or SWM);
  * Monoclonal B cell lymphocytosis (MBL);
  * Early stage asymptomatic low-grade lymphomas; or
  * Other precursor conditions or clonal genetic abnormalities of the blood/bone marrow that do not meet criteria for symptomatic hematological malignancy, or patients exposed to prior chemotherapies (e. g., alkylating agents, platinum derivatives, taxanes, topo-2 inhibitors, anti-metabolites, systemic radioisotopes).
* Patients must be at least 18 years of age to participate in this research.
* Inclusion of Women and Minorities -- In accordance with NIH guidelines, women and members of minority groups and their subpopulations will be included in this protocol.

Exclusion Criteria:

* Patients with Known or Suspected Precursor Hematological Cancer are NOT EXCLUDED
* Evidence of symptomatic or active hematological malignancy. Patients enrolled on clinical trials for precursor diseases are NOT excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Known or Suspected Precursor Hematological Cancer
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Identify molecular changes in cells of patients with precursor hematological malignancies | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute at St. Elizabeth's, Brighton, Massachusetts
  - Dana Farber Cancer Institute at Merrimack Valley, Methuen, Massachusetts
  - Dana Farber Cancer Institute at Milford Regional Medical Center, Milford, Massachusetts
  - Dana Farber Cancer Institute at South Shore, Weymouth, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Dana Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire